CLINICAL TRIAL: NCT03590132
Title: A Dual Inoculation Approach to Alcohol Prevention Among African American Youth
Brief Title: Strong African American Families STEPS Project
Acronym: SAAF-STEPS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Georgia (Other)
Responsible Party: Principal Investigator, Steve Kogan, Professor, University of Georgia
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Prevention
Other Study IDs: UGA045608
Record Dates: First submitted 2018-06-12; First posted 2018-07-18 (Actual); Last update posted 2019-06-19 (Actual); Status verified 2019-06

CONDITIONS: Adolescent Alcohol Use
Keywords: adolescent; alcohol; family-centered prevention; African American
MeSH Terms: conditions — Underage Drinking

STUDY DESIGN:
Intervention Model Description: A 4 arm trial, participants receive either a preadolescent intervention only, a mid-adolescent intervention only, both preadolescent and mid-adolescent intervention, or no intervention
Who Masked: Care Provider, Outcomes Assessor
Masking Description: Neither the interventionists or the assessors were given information on participants' treatment group; however there is only partial masking for providers given that attendance in the program suggests some information on experimental group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- SAAF (Experimental): participants in this arm receive the SAAF intervention at age 11-12.
  Interventions: Behavioral: Strong African American Families Program
- SAAF-T (Experimental): participants in this arm receive the SAAF-Teen intervention at age 14-15.
  Interventions: Behavioral: Strong African American Families--Teen Program
- SAAF SAAF-T (Experimental): participants in this arm receive SAAF at age 11-12 and later receive SAAF-Teen at age 14-15
  Interventions: Behavioral: Strong African American Families Program; Behavioral: Strong African American Families--Teen Program
- Control (No Intervention): These participants receive no interventions.

INTERVENTIONS:
Behavioral: Strong African American Families Program — SAAF is a 7 session family skills training program
  Other Names: SAAF
  Arms: SAAF; SAAF SAAF-T
Behavioral: Strong African American Families--Teen Program — SAAF-T is a 5 session family skills training program
  Other Names: SAAF--T
  Arms: SAAF SAAF-T; SAAF-T

SUMMARY:
The most common approach to preventing alcohol use involves providing a well-designed program in preadolescence just prior to or upon entering middle school. This approach does not have long-lasting effects or address the risk factors that lead many youth to use alcohol in high school. This study tested a strategy that compares offering effective programs at the transition to middle school and the transition to high school with only offering a program at either one of the transitions or no programs at all.

DETAILED DESCRIPTION:
Alcohol use is a leading cause of morbidity and mortality among high school students. Annually, underage drinking leads to more than 3,000 deaths and 2.6 million other harmful events, resulting in $5.4 billion in medical costs, $14.9 billion in work loss and other resource costs, and $41.6 billion in lost quality of life. This public health crisis has engendered considerable attention from prevention scientists, who have specified guidelines for the development of primary prevention programs and the timing of their implementation. The present research is based on critical limitations in the prevailing model for implementing primary prevention for alcohol use. This model focuses on delaying alcohol use onset among youth who begin use in middle school (ages 11-14). Based on studies that linked early use to a high-risk behavioral trajectory in adolescence, prevention scientists translated data on risk and protective processes for early-onset alcohol use into primary prevention programs for youth to be implemented during or just prior to the transition to adolescence. This model has informed numerous randomized prevention trials and investigations of prevention implementation. An unquestioned premise of this model involves the adequacy of a single preadolescent "inoculation" of prevention programming to protect youth into the high school years.

The proposed trial addresses empirical and theoretical limitations to the preadolescent/single inoculation paradigm. First, inclusive reviews reveal that primary prevention programs implemented in early adolescence fail to achieve robust, long-term results. Second, studies of alcohol use trajectories reveal patterns of onset in high school with rapid escalation that culminate in high levels of alcohol use. Third, in the prevailing paradigm, targeting early adolescent risk processes is assumed to be sufficient to equip youth for the novel risk processes they will encounter in high school. In contrast, this study investigates the proposition that achievement of public health impact requires a "dual-inoculation" prevention strategy, one that addresses both onset in early adolescence and mid-adolescence and provides developmentally tailored curricula at each transition.

Based on longitudinal studies with rural African American families that documented the changing context of alcohol use risk and protective processes from late childhood through adolescence, scientists at the Center for Family Research developed a series of developmentally appropriate, family-centered preventive interventions that have proven efficacious in in preventing alcohol use: the Strong African American Families (SAAF) program for youth age 10-12 and the SAAF-Teen program for youth age 14-16. These programs afford a unique opportunity to test dual-inoculation hypotheses. Unlike medical inoculations of a vaccine, it is not appropriate to give the same inoculation to an 11-year-old that one gives a 14-year-old. Rather, each preventive inoculation must be tailored to address the most salient risk and protective processes at particular developmental transitions.

This study will recruit a sample of 460 African American families into a four-arm randomized prevention trial and evaluate the differential alcohol prevention effects of (a) a dual inoculation of prevention (youth receive SAAF at age 11 and SAAF-Teen at age 14) compared with (b) receipt of a preadolescent inoculation (SAAF at age 11), (c) receipt of a mid-adolescent inoculation (SAAF-Teen at age 14), or (d) a minimal contact control.

Specific efficacy aims are to:

1. Test the hypothesis that rural African American youth randomly assigned to participate in two prevention inoculations will demonstrate lower rates of alcohol use initiation, frequency of use, binge drinking, and alcohol-related problems in high school than will youth who receive a preadolescent inoculation only, a mid-adolescent inoculation only, or no inoculations.
2. Investigate the intervening processes that account for the relative efficacy of a dual inoculation. Specifically, we expect that intervention-targeted early adolescent protective processes, early adolescent alcohol use outcomes, and intervention-targeted mid-adolescent protective processes will account for group differences in alcohol use in high school.

   To facilitate the potential dissemination of a dual inoculation approach, this study investigates the cost-effectiveness of a dual inoculation relative to preadolescent, mid-adolescent, or control conditions.

   The specific cost-effectiveness aim is to:
3. Conduct a cost-effectiveness analyses that estimates the incremental cost of a dual inoculation compared to single inoculations and no inoculations per additional unit decrease in alcohol use initiation, escalation, binge drinking, and alcohol-related problems. This study will investigate an ancillary hypothesis involving the incremental cost difference per outcome unit between preadolescent and mid-adolescent inoculations relative to the control condition.

ELIGIBILITY:
Inclusion Criteria:

* self reported African American
* 5th grade

Exclusion Criteria:

* unable to attend a family-centered prevention intervention due to incapacitation of youth
* unable to attend a family-centered prevention intervention due to incapacitation of youth

Ages: 11 Years to 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 472 (Actual)
Dates: Start 2012-12-10 (Actual); Primary Completion 2018-11-30 (Actual); Study Completion 2018-11-30 (Actual)

PRIMARY OUTCOMES:
Alcohol use in past 3 months (single item) | 3 months
  Youth complete this single item from Monitoring the Future Study assessing the frequency of alcohol use in the past 3 months. There is an ordinal response scale ranging from 0 (none) to 6 (30 or more times). Higher response numbers indicate a worse outcome (more alcohol use).
Frequency of cannabis use in the past 3 months (single item) | 3 months
  Single item from Monitoring the Future Study assessing frequency of marijuana use in the past 3 months. There is an ordinal response scale ranging from 0 (none) to 6 (30 or more times). Higher responses indicate a worse outcome (more marijuana use in the past 3 months).
Monitoring the Future: Total substance use (summative index of use of alcohol, cannabis, and nicotine) | 3 months
  Youth complete 3 single items from the Monitoring the Future study indexing the frequency of their use of alcohol, cannabis, and nicotine in past 3 months. There is an ordinal response scale ranging from 0 (none) to 6 (30 or more times) for each item. The three items are summed yielding a scale ranging from 0-18. Higher response numbers indicate a worse outcome (more substance use).

SECONDARY OUTCOMES:
Center for Epidemiological studies-Depression scale | Past 7 days
  Parent complete this 20 item measure of depressive symptoms. Responses to each item are on a scale from 0 to 3; responses are summed. Items are summed. Scores range from 0-60 with higher scores indicate more depressive symptoms in the past week (a worse outcome).
The National Survey of Adolescents Conduct Problems Subscale | past 3 months
  Youth complete a 15 Item scale from the National Survey of Adolescents which refer to different conduct problems. Youth provide the number of times they enacted each behavior in the past 3 months. These responses are summed. Scores can range from 0-99 with higher scores indicating more engagement in conduct problems.
Center for Epidemiological Studies-Depression Scale-Child Version | past 7 days
  Youth complete this 20 item measure of depressive symptoms. Responses to each item are on a likert scale from 0 to 3; responses are summed. Scores range from 0-60 with higher scores indicate more depressive symptoms in the past week (a worse outcome).

IPD SHARING:
Plan to Share IPD: No
Participants have not consented to data being shared outside of research team

REFERENCES:
- [Derived] Kogan SM, Reck AJ, Tiwari B, Thapha JR, Carter S, Oshri A, Koss K, Ahn SJ, Beach S, Fisher S, Smith E, Zhang L. Family-Centered Prevention Attenuates the Association Between Structural Racism Risk and Black Adolescents' Low Self-regulation and Externalizing Behaviors: Secondary Analysis of a Randomized Clinical Trial. Prev Sci. 2025 Aug;26(6):932-942. doi: 10.1007/s11121-025-01828-5. Epub 2025 Jul 17. PMID 40676489
- [Derived] Kogan SM, Kwon E, Brody GH, Azarmehr R, Reck AJ, Anderson T, Sperr M. Family-Centered Prevention to Reduce Discrimination-Related Depressive Symptoms Among Black Adolescents: Secondary Analysis of a Randomized Clinical Trial. JAMA Netw Open. 2023 Nov 1;6(11):e2340567. doi: 10.1001/jamanetworkopen.2023.40567. PMID 37910105